CLINICAL TRIAL: NCT05455099
Title: Multicenter Study of Carotid Artery Ultrafast Pulse Wave Velocity (UFPWV) in Obese Adults
Brief Title: A Multicenter Study of Ultrafast Pulse Wave Velocity in Obese Chinese Han Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Other Study IDs: CO-UFPWV-01
Record Dates: First submitted 2022-07-06; First posted 2022-07-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Carotid Artery Diseases
Keywords: Obesity; Pulse Wave Velocity; Carotid Artery Diseases; Cerebrovascular Disorders; Vascular Diseases; Cardiovascular Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases
MeSH Terms: conditions — Carotid Artery Diseases; Obesity; Cerebrovascular Disorders; Vascular Diseases; Cardiovascular Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese group: Participants will be assigned to obese group (body mass index 24.0-27.9 kg/m²). Based on the inclusion criteria, 1200 overweight Han people（body mass index 24.0-27.9 kg/m²）and both sexes will be recruited in the analysis. The values of ultrafast pulse wave velocity will be obtained.
  Interventions: Radiation: Carotid ultrasound examination 1
- overweight group: Participants will be assigned to overweight group (body mass index ≥ 28.0 kg/m²). Based on the inclusion criteria, 1200 obese Han people（body mass index ≥28.0 kg/m²） and both sexes will be recruited in the analysis. The values of ultrafast pulse wave velocity will be obtained.
  Interventions: Radiation: Carotid ultrasound examination 2

INTERVENTIONS:
Radiation: Carotid ultrasound examination 1 — Participants will be assigned to obese group (body mass index 24.0-27.9 kg/m²). Carotid pulse wave velocity of all participants were measured by ultrafast ultrasound imaging technology using SuperSonic Imagine's explorer ultrasound system.
  Groups: obese group
Radiation: Carotid ultrasound examination 2 — Based on the inclusion criteria, 1200 overweight Han people（body mass index ≥28.0 kg/m²） and both sexes will be recruited in the analysis. The values of ultrafast pulse wave velocity will be obtained.
  Groups: overweight group

SUMMARY:
Ultrafast pulse wave velocity (UFPWV) is a novel non-invasive method developed recently to evaluate pulse wave velocity (PWV). This multi-center clinical trial aims to evaluate the feasibility of UFPWV in the evaluation of the carotid stiffness of overweight and obese population and investigate the correlation between overweight/obesity and subclinical atherosclerosis, providing an important theoretical basis for early monitoring and risk assessment of carotid atherosclerosis in overweight/obese people.

DETAILED DESCRIPTION:
In recent years, with the change of people's lifestyle and dietary structure, overweight and obesity have become serious problems threatening public health. During 1975-2016, the worldwide prevalence of overweight and obesity increased year by year. By 2016, about 40% of adults were overweight and obese, of which 2.3% of men and 5.0% of women were severely obese (i.e. body mass index ≥ 35 kg/m²). The number of overweight and obese people in China is growing rapidly. Report on the Nutrition and Chronic Disease Status of Chinese Residents (2020 version) shows that over 50% Chinese obese adults have overweight and obesity. Overweight and obesity have become one of the most serious public health problems in China. Previous studies have found that overweight and obesity are often accompanied by abnormalities of blood glucose, blood pressure and blood lipids, leading to dysfunction of vascular endothelial cells and changes in the structure and function of vascular wall, which are closely related to atherosclerosis. Therefore, early detection of atherosclerosis and timely intervention measures can effectively prevent and reduce the occurrence and development of atherosclerosis.

At present, carotid intima-media thickness (CIMT) can be clinically used to evaluate carotid atherosclerosis, which can evaluate the morphological changes of carotid artery, but it cannot be used to evaluate the stiffness of carotid artery. PWV is the gold standard for evaluating arterial stiffness. However, the conventional PWV measurement method can evaluate the stiffness of long-distance artery. Evaluated outcomes are affected by height and body mass, and therefore, the evaluation accuracy of PWV can be limited.

UFPWV is a novel noninvasive method developed in recent years to evaluate PWV. It can be used to evaluate PWV of local artery. Different from the conventional PWV method, UFPWV has a very high frame rate, up to 2000 frames/s, and can track the movement of arterial wall at specific segments in real time. UFPWV can obtain PWV at the beginning and end of systole by tracking and automatic analysis. In recent years, increasing attention has been paid to the role of UFPWV in the evaluation of carotid artery. UFPWV has been used in the study of carotid arteries in normal people, vascular Ehlers-Danlos syndrome, hypertension, hyperlipidemia, diabetes and other groups.

In the early stage, First Hospital of China Medical University participated in the national multi- center, large-sample trial: multi-center study on normal value of ultrafast pulse wave velocity in Chinese Han adults. The center has accumulated rich experience during the project implementation. The center determined the normal reference value of UFPWV for Chinese Han adults and verified that UFPWV has good measurement repeatability. At the same time, the project team had applied UFPWV technology to study early carotid atherosclerosis in patients with metabolic syndrome and coronary slow flow phenomenon. The results show that UFPWV has been accelerated without marked thickening of CIMT, which preliminarily proves that UFPWV can accurately and sensitively detect early carotid atherosclerosis.

This study aims to evaluate the feasibility of UFPWV in carotid stiffness of overweight and obese people, and correlate overweight/obesity with subclinical atherosclerosis, so as to provide an important theoretical basis for early monitoring and risk assessment of carotid atherosclerosis in overweight/obese people.

ELIGIBILITY:
Inclusion Criteria:

* Han nationality;
* Age ≥18 - 80 years;
* Body mass index ≥ 24 kg/m²;
* Blood pressure ≥ 90/60 mmHg (1 mmHg = 0.133 kPa);
* Fasting blood glucose level ≥ 3.9 mmol/L;
* No abnormality in cardiovascular and respiratory system found by physical examination;
* Normal findings in routine blood test, routine urine test, liver function and kidney function;
* No history of cardiovascular disease, respiratory system disease, liver and kidney disease except hypertension, diabetes or hyperlipidemia;
* Electrocardiogram examination showed no arrhythmia or myocardial infarction;
* No structural cardiac abnormalities (such as moderate or above cardiac valve regurgitation, abnormal ventricular wall motion, congenital heart disease, cardiomyopathy, pericardial lesions) were found by echocardiography, and left ventricular ejection fraction ≥ 53%;
* No marked abnormality in ultrasonography of the liver, gallbladder, pancreas, spleen and kidney;
* Normal findings in carotid ultrasound examination.

Exclusion Criteria:

* Hepatorenal insufficiency;
* Respiratory diseases: Acute or chronic respiratory diseases;
* Large artery diseases: aortic dilatation, aortic dissection, aortic coarctation, multiple Takayasu arteritis, etc;
* Special diseases: history of malignant tumor, acute or chronic infection, moderate to severe anemia, disability or mental disorder, autoimmune diseases, acquired immunodeficiency syndrome, etc;
* Pregnant or lactating women;
* Recent history of surgery and trauma;
* Organ transplant;
* Poor ultrasonic image quality, which cannot meet analysis requirement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population description * (only for observational study): 2400 overweight or obese adults will be recruited from physical examination center. They will be assigned to overweight group (body mass index 24.0-27.9 kg/m²; n = 1200) and obese group (body mass index ≥ 28.0 kg/m²; n = 1200).
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity（m/s）at the ending of the systole (ES) of carotid artery | 1 day after admission
  To evaluate the pulse wave velocity（m/s）at the ending of the systole (ES) of carotid artery in overweight/obese population.

SECONDARY OUTCOMES:
Pulse wave velocity（m/s）at the beginning of the systole (BS) of carotid artery | 1 day after admission
  To evaluate the pulse wave velocity（m/s）at the beginning of the systole (BS) of carotid artery in overweight/obese population
Carotid artery intima-media thickness (IMT) | 1 day after admission
  IMT（mm） reflects the change of vascular wall structure, which is used to evaluate early atherosclerosis.
Serum biochemical index | 1 day after admission
  Serum laboratory testing for blood total cholesterol level in mmol/L, high-density lipoprotein level in mmol/L, low-density lipoproteins level in mmol/L, triglycerides level in mmol/L, and fasting blood-glucose level in mmol/L will be examen.

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Ma, Ph.D, Principal Investigator — the First Hospital of China Medical Univeristy
Locations (22):
- China (22):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Guangdong Province Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - the Fifth Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hebei General Hospital, Shijiazhuang, Hebei
  - the First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xiangyang No.1 Peoples Hospital, Xiangyang, Hubei
  - Affiliated Hospital of Nanjing University of Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Province Official Hospital, Nanjing, Jiangsu
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - the First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Affiliated Central Hospital of Shenyang Medical College, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Xi'an Daxing Hospital, Xi'an, Shaanxi
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Yuechi People's Hospital, Guang’an, Sichuan
  - People's Hospital of Leshan, Leshan, Sichuan
  - Jiangyou People's Hospital, Mianyang, Sichuan
  - NHC Key Laboratory of Hormones and Development, CHU Hsien-i Memorial Hospital and Tianjin Institute of Endocrinology, Tianjin, Tianjin Municipality
  - Gejiu People's Hospital, Gejiu, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided